CLINICAL TRIAL: NCT04829630
Title: Immunity Persistence After Abridged Intradermal Rabies PEP
Acronym: RESIST-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur du Cambodge (Other); Institut Pasteur de Madagascar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-064
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2021-11

CONDITIONS: Rabies
Keywords: rabies; vaccine; Post-exposure prophylaxis; Persistent immunity; Short protocol
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: * 90 subjects in Cambodia or Madagascar who received ID PEP by 3 sessions/1 week at least two (30 subjects), five (30 subjects) or 10 years earlier (30 subjects),
  * 90 subjects in Cambodia or Madagascar who received ID PEP by 4 sessions/1 month at least two (30 subjects), five (30 subjects) or 10 years earlier (30 subjects),
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subjects who received three vs. four ID PEP at least two, five or 10 years earlier (Other): * 30 subjects who received three ID PEP at least two years earlier in Cambodia
  * 30 subjects who received three ID PEP at least five years earlier in Cambodia
  * 30 subjects who received three ID PEP at least 10 years earlier in Cambodia
  * 30 subjects who received four ID PEP at least two years earlier in Madagascar
  * 30 subjects who received four ID PEP at least five years earlier in Madagascar
  * 30 subjects who received four ID PEP at least 10 years earlier in Madagascar
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — * day 0 : questionnaire, blood sampling and vaccine booster (a single session of two intradermal doses of 0.1 mL)
  * day 7 : questionnaire and blood sampling

SUMMARY:
After exposure, rabies can be prevented in almost 100% of cases by the administration of sufficient and timely post-exposure prophylaxis (PEP). PEP is based on wound cleansing, antisepsis, administration of rabies vaccine as well as rabies immunoglobulin, if reviewed. However, anti-rabies PEP remains too often out of financial and / or geographic access, especially for poor and / or rural populations in endemic countries who remain the most exposed to the risk of contracting rabies. Two major studies planned in Cambodia between 2014 and 2018 - the RESIST 0/1 clinical - epidemiological study and the RESIST-2 study on the antibody response to the vaccine - provided the basis that allowed a change in international recommendations on PPE. Since April 2018, the new "IPC protocol" of three sessions of reduced double doses (0.1 mL x 2) administered intradermally (ID) over one week has replaced the already very effective "TRC protocol" of four sessions over one month which was the reference dose-sparing protocol for endemic countries until 2018. It remains to be determined whether the IPC protocol (3 sessions / 1 week) confers long-term immunity equivalent to that obtained after a TRC ID protocol (4 sessions / 1 month). This question is of importance to public health decision-makers and clinical teams in endemic countries who would hesitate to switch to the abbreviated IPC protocol.

DETAILED DESCRIPTION:
This is a multicenter, randomized, non-inferior clinical trial with samples for examinations and vaccination booster.

To achieve this study, persons who previously received PEP and of any age (including children), gender or medical condition (including pregnant women) and whichever the status of the dog which bit at least 2, 5 or 10 years ago will be contacted and invited to participate to the study.

This study will take place in two centers :

* The rabies prevention center at Institut Pasteur du Cambodge
* The rabies prevention center at Institut Pasteur de Madagascar. The study will be coordinated by Institut Pasteur in Paris which will subsequently conduct the analysis in collaboration with researchers at Institut Pasteur du Cambodge and Institut Pasteur de Madagascar.

This study will take place in two visits :

* the first visit (day 0) : after receiving consent from the participants, the member of the investigating team will perform the blood sample, followed by a single session of two intradermal doses of 0.1 mL. The investigators will also carry out measurements and complete the questionnaire with the participant.
* the second visit (day 7) : a follow-up visit will be performed by a member of the investigating team who will perform a second blood sample to all the participants to the study. The investigator will complete a second paper CRF with the participants to document any unwanted effects which may have occurred during the seven days between the inclusion visit and the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* person Identified in IP Cambodia or IP Madagascar records for having received ID PEP by 4 sessions/1 month or 3 sessions/1 week at least two, five or 10 years earlier, with no rabies boosting since that time;
* person Who received information adapter to his/her age and who signed the consent form (or his/her legal tutors)

Exclusion Criteria:

* person who received Rabies vaccine booster since the earlier PEP
* person with allergy or other severe unwanted effect at the time of the earlier PEP

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Antibody titers measured (FAVN, RFFIT) and cellular immunity markers one week after a single session of ID rabies vaccine boosting in the two groups | 1 year
  Absence of statistically significant difference between antibody titers Fluorescent Antibody Virus Neutralization test (FAVN) and Rapid Fluorescent Foci Inhibition Test (RFFIT) and cellular immunity markers one week after a single session of ID rabies vaccine boosting in persons who have received a 3 sessions/1 week vs. 4 sessions/ 1 month ID PEP at least 2, 5 or 10 years earlier.

SECONDARY OUTCOMES:
Antibody titers measured by FAVN and RFFIT and immune response before a single session of ID rabies vaccine boosting in the two groups | 1 year
  Equivalence of antibody titers and immune response before a single session of ID rabies vaccine boosting in persons who have received a 3 sessions/1 week vs. 4 sessions/ 1 month ID PEP at least 2, 5 or 10 years earlier.
Antibody titers measured by FAVN and RFFIT in all subjects for comparison | 1 year
  Equivalence of antibody titers measured using FAVN compared to the RFFIT used as reference.

CONTACTS AND LOCATIONS:
Overall Officials: Perrine Parize, MD, Study Director — Institut Pasteur
Locations (2):
- Institut Pasteur du Cambodge, Phnom Penh, Cambodia
- Institut Pasteur de Madagascar, Antananarivo, Madagascar